CLINICAL TRIAL: NCT04364659
Title: Targeting Inhibitory Control Using Computerised Training Among Patients With Bulimia Nervosa and Binge Eating Disorder
Brief Title: Computerised Training for Binge-Subtype Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS ID: 252717
Record Dates: First submitted 2020-03-09; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-10

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food-specific ICT + TAU (Experimental): Participants in the Food-specific ICT + TAU group will be encouraged to complete the FoodT phone app (a food-specific go/no-go task) and a food diary daily for four weeks. After four weeks, they will be asked to complete a post-intervention questionnaire. After eight weeks, they will be asked to complete a follow-up questionnaire.
  Interventions: Behavioral: Food-Specific Inhibitory Control Training (FoodT App)
- TAU (No Intervention): Participants in the TAU group will not receive the Food-specific ICT. After four weeks, they will be asked to complete a 'post-intervention' questionnaire. After eight weeks, they will be asked to complete a follow-up questionnaire.

INTERVENTIONS:
Behavioral: Food-Specific Inhibitory Control Training (FoodT App) — FoodTrainer (FoodT) is a simple game that aims to train individuals to 'stop' to certain unhealthy foods. Repeatedly playing this game is hypothesised to help build associations between certain foods (such as chocolate) and stopping, putting the brakes on unhelpful eating behaviour.
  Arms: Food-specific ICT + TAU

SUMMARY:
This research project aims to explore the feasibility of a computerised training to reduce approach to high energy-dense foods among individuals who binge eat. The computerised intervention used will be an inhibitory control training, particularly, a food-specific go/no-go task. Eighty adults with a diagnosis of bulimia nervosa or binge eating disorder who are currently receiving psychological and/or pharmacological treatment for their eating disorder will be recruited and randomised to receive the computerised training in addition to treatment as usual (experimental group: training + TAU) or treatment as usual only (control group: TAU). Participants will complete questionnaires at baseline (T0), post-intervention (T1; 4 weeks), and follow-up (T2; 8 weeks).

Participants will be asked to complete the computerised training for 4 weeks using a mobile app called FoodT. The computerised training consists of completing a food-specific go/no-go task to reduce approach to high energy-dense foods.

The results of this study will build steps for future larger-scale interventions and improve understanding of psychological mechanisms involved in binge eating behaviour.

DETAILED DESCRIPTION:
Participants will learn about the study through flyers, e-mail, and social media (i.e. Facebook and twitter), which will describe the main eligibility criteria and the researcher's contact information. Participants will also learn about the study from their eating disorder unit if they are currently outpatients at one of the identification centres. Inpatients will not be recruited.

Interested individuals will be asked to contact the researchers, who will then send an information sheet detailing the study procedure and what participation would involve. After reading the information sheet, interested individuals will be contacted by the researchers in order to confirm all eligibility criteria including diagnostic assessment. If these are met, a PDF of the consent form will be sent to the participants, including information about their rights as participants and their ability to withdraw at any time without having to give a reason. Participants who sign the consent form will respond to the e-mail with the attached document. Next, participants will be randomly allocated to the experimental condition (TAU + training) or control group (TAU only). Researchers will then inform the participant which group they have been allocated to. If they are in the intervention group, the researcher will contact the participant to give details about the training. All participants will be asked to complete a battery of questionnaires on Qualtrics, an online platform.

The questionnaires will collect data regarding: 1) a demographic information, 2) eating disorder symptoms (Eating Disorders Examination Questionnaire; Self-Regulation of Eating Behaviour Questionnaire; Adult Eating Behaviour Questionnaire; Yale Food Addiction Scale; Food Liking Task), 3) impulsivity (Negative Urgency Scale), 4) symptoms of anxiety or depression (GAD-7 anxiety; PHQ-9 Depression) and 5) quality of life (EQ-5D-3L).

Participants in the intervention group will be asked to complete the training and a food diary for four weeks. After the four weeks, all participants will be asked to complete the same battery of questionnaires (except for the demographic questionnaire). One month post-intervention, a follow-up questionnaire will also be sent.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of bulimia nervosa or binge eating disorder
2. Age 18-60 years old

2) BMI ≥ 18.5 3) Fluency in English

Exclusion criteria:

1. A diagnosis of psychosis
2. A visual impairment that cannot be corrected by glasses or lenses
3. Cognitive or neurological impairment
4. Drug or alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | At 4 weeks.
  Feasibility as defined by: 1) the recruitment of 75% of the target number (N = 80), 2) participants' adherence to the training task, with ≥ 75% of participants completing at least 8 training sessions, and 3) participants' retention in treatment, with ≥ 80% of the sample completing the end of training measures.
Acceptability of intervention | Feedback forms will be completed 8 weeks post-randomisation (at follow-up).
  Feedback forms will be used to assess the acceptability of the training, including participants' view of the helpfulness, practicality, and potential improvements to it.
Acceptability of intervention | Focus groups will be conduced 2 weeks after recruitment has ended.
  Focus groups will be used to assess the acceptability of the training, including participants' view of the helpfulness, practicality, and potential improvements to it.
Efficacy: Changes in Binge Eating Frequency | Measured at baseline, at 4 weeks, and at 8 weeks (follow-up).
  The primary outcome aim is to examine the efficacy of app-based food-specific go/no-go training in targeting binge-eating frequency (as measured using item #13 on the Eating Disorder Examination Questionnaire). It is hypothesised that participants would exhibit reductions in binge eating frequency, with stronger effects in the experimental group (training + TAU) compared to the control (TAU) group. Participants are free to enter any numerical value, with a greater value indicating a higher frequency of binge eating.

SECONDARY OUTCOMES:
Efficacy: Changes in Eating Disorder Psychopathology | Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this secondary outcome is to examine the efficacy of app-based food-specific go/no-go training in targeting eating disorder psychopathology (as measured using the Global Eating Disorder Examination Questionnaire score). It is hypothesised that participants will exhibit reductions in these outcomes, with stronger effects in the experimental group (training + TAU) compared to the control (TAU) group. The mean score can range from 0-6, with higher scores indicating higher eating disorder psychopathology.
Efficacy: Changes in High Energy-Dense Food Valuation | Measured at baseline, at 4 weeks (post-intervention), Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this secondary outcome is to examine the efficacy of app-based food-specific go/no-go training in targeting high energy-dense food valuation (as measured using the Food Rating Test). It is hypothesised that participants will exhibit reductions in these outcomes, with stronger effects in the experimental group (training + TAU) compared to the control (TAU) group. The mean score can range from 0-100, with higher scores indicating greater high energy-dense food valuation.
Efficacy: Changes in Food Approach | Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this secondary outcome is to examine the efficacy of app-based food-specific go/no-go training in targeting food approach (as measured using the Adult Eating Behaviour Questionnaire, food approach sub scale). It is hypothesised that participants will exhibit reductions in these outcomes, with stronger effects in the experimental group (training + TAU) compared to the control (TAU) group. Participant responses range from 1-5, ranging from strongly disagree to strongly agree. Higher scores indicate greater food approach behaviour.
Efficacy: Changes in Food Addiction | Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this secondary outcome is to examine the efficacy of app-based food-specific go/no-go training in targeting food addiction (as measured using the Yale Food Addiction Scale). It is hypothesised that participants will exhibit reductions in these outcomes, with stronger effects in the experimental group (training + TAU) compared to the control (TAU) group. The mean score can range from 0-4, with higher scores indicating greater food addiction.

OTHER OUTCOMES:
Exploratory: Changes in Depression | Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this experimental outcome is to explore whether individuals in the experimental group (training + TAU) will show reductions in depression (as measured using the Patient Health Questionnaire- 9), and if so, whether the reduction is greater than that found among participants in the control group (TAU). The total score can range from 0-27, with greater scores indicating greater levels of depression.
Exploratory: Changes in Anxiety | Measured at baseline, at 4 weeks (post-intervention), and at 8 weeks (follow-up).
  The aim of this experimental outcome is to explore whether individuals in the experimental group (training + TAU) will show reductions in anxiety (as measured by the Generalised Anxiety Disorder-7), and if so, whether the reduction is greater than that found among participants in the control group (TAU). The total score can range from 0-21, with higher scores indicating greater levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Treasure, OBE, PhD, FRCP, FRCPsych, Principal Investigator — Institute of Psychiatry, Psychology, & Neuroscience, King's College London; Valentina Cardi, PhD, Study Director — Institute of Psychiatry, Psychology, & Neuroscience, King's College London; Natalia Lawrence, PhD, Study Chair — University of Exeter; Johanna Keeler, BSc, Study Chair — University of Exeter
Locations (1):
- King's College London, London, United Kingdom